CLINICAL TRIAL: NCT07000734
Title: Fortifying Healthy Behaviors, Optimizing Medical Therapies and Enhancing Cognitive Function in Older Adults-pilot Study
Acronym: FOES
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202503023
Record Dates: First submitted 2025-05-19; First posted 2025-06-03 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Aging; Cognitive Decline; Older Adults; Cardiovascular; Sedentary Behaviors; Immune Senescence; Motor Function
MeSH Terms: conditions — Cognitive Dysfunction; Sedentary Behavior | interventions — Dasatinib; Quercetin; Dietary Supplements; Vortioxetine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Behavioral lifestyle management plus dasatinib, quercetin and vortioxetine (Experimental): Open label multicomponent, personalized intervention incorporating behavioral and medicinal therapies
  Interventions: Behavioral: Risk managment; Drug: Dasatinib; Dietary Supplement: Quercetin (dietary supplement); Drug: Vortioxetine

INTERVENTIONS:
Behavioral: Risk managment — Behavioral lifestyle changes including an exercise program, healthy eating recommendations, reviewing medical management for cardiometabolic risk conditions, deprescribing review for brain toxic meds, online cognitive training, as well as recommendations to improve sleep quality, or smoking cessation as needed
Drug: Dasatinib — dasatinib 100mg The intervention will involve the participant taking dasatinib 100mg and quercetin 1250ng combined, intermittenly throughout the trial
  Other Names: sprycel; sophoretin
Dietary Supplement: Quercetin (dietary supplement) — e intervention will involve the participant taking dasatinib 100mg and quercetin 1250ng combined, intermittenly throughout the trial
  Other Names: quercetine; Vitamin P
Drug: Vortioxetine — Participants will be prescribed vortioxetine to take daily, in combination with online cognitive training
  Other Names: Trintellix; Brintellix

SUMMARY:
The purpose of this research study is to explore ways to improve motor, cognitive and immune functions for aging adults using multiple techniques like lifestyle changes and risk factor management, as well as medications and supplements believed to have a positive effect on health.

DETAILED DESCRIPTION:
The goal in this pilot open-label study is to conduct a feasibility test of a multi-component, personalized intervention designed to improve the aging human healthspan. The trial will recruit at least 20 adults aged 50-70, both male and female. The total time of study participation is up to 5 months.

The intervention will last for approximately 3 months, with testing of motor, cognitive, and immune outcomes before and after the intervention.

The intervention consist of three components:

1. Fortify Healthy Behaviors: behavioral lifestyle management that combines an exercise program, healthy eating behaviors and optimizing sleep quality;
2. Optimize Medical Therapies: reviewing the participants cardiovascular risk factors, smoking cessation when indicated, treatment with the senolytic medication dasatinib combined with the antioxidant quercetin , and dietary supplements relevant for brain, bone and immune system functioning; and
3. Enhance Cognitive Function: vortioxetine (an antidepressant shown to have pro-cognitive properties), in combination with digital cognitive training to improve fluid cognition and memory, and deprescribing of drugs with CNS toxicity (i.e. those that cause cognitive difficulties).

The outcome assessments will be measured both pre- and post-intervention and up to three times at each time point. These assessments will look at biomarkers related to aging. Assessments will include strength and endurance tests, validated neuropsychological tests, and a blood drawn to look at immune function.

An MRI scan will also be offered to participants who are able to undergo the scan to look at brain health and aging, both pre- and post-intervention.

ELIGIBILITY:
Participants must be residents of Illinois or Missouri and able to come to St. Louis offices in person.

Inclusion Criteria:

* Ages 50-70
* Able to come to the research center for testing and intervention visits.
* Sedentary (no moderate exercise and no more than 15-minutes per day of light exercise (confirmed via interview with participants)).
* BMI≥27 or Body Roundness index ≥6
* Able to provide informed consent.

Exclusion Criteria:

* Dementia or other clinical neurodegenerative illness (e.g., Parkinson's disease, cerebrovascular disease unless minor eg one lacunar infarct with minimal/no impairment) per self-report or medical records.
* Medical conditions that suggest shortened lifespan (such as metastatic cancer), severe/uncontrolled psychiatric disorders or conditions that would prohibit safe participation.
* Unable to perform study assessments.
* Alcohol or substance abuse within 6 months per self-report or medical records.
* Concurrent cognitive training, such as brain-training software, or other interventions expected to affect neuroplasticity.
* Any drug that interacts pharmacokinetically, or is contraindicated with study interventions (examples would include high-dose SSRI that should not be combined with vortioxetine)
* PI has discretion to exclude potential participants eg if their health status appears either too good or too poor to be amenable to intervention

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-07-28 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Number of participants who completed the outcome measure assessments and intervention | 5 months
  Reviewing feasibility outcomes including recruitment, retention, participant adherence, interventionist fidelity to behavioral treament protocols and collection of outcome measures.

OTHER OUTCOMES:
Motor function | 5 months
  Endurance capacity; 6 Minute Walking Test Lower body power: Leg dynamometer Skeletal muscle: D3 creatine dilution
Cognitive Function | 5 months
  NIH Toolbox Cognitive Battery, Fluid Cognition Composite. Each of the 5 subscales have a mean of 100 with a standard deviation of 15.
Immune Function | 5 months
  Blood draws to look at biomarkers related to immune function

CONTACTS AND LOCATIONS:
Overall Officials: Eric Lenze, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
Contact PI